CLINICAL TRIAL: NCT00920985
Title: Multi-Center, Double-Blind, Double-Dummy, Randomized, Parallel-Group Study to Evaluate Cycle Control, Bleeding Pattern, Blood Pressure, Lipid and Carbohydrate Metabolism of the Transdermal Contraceptive Patch (Material no. 80876395 / 2.1 mg Gestodene and 0.55 mg Ethinylestradiol) Versus an Oral Comparator Containing 20 µg Ethinylestradiol and 100 µg Levonorgestrel in a 21-day Regimen for 7 Cycles in 400 Women
Brief Title: US Cycle Control and Blood Pressure Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 91556
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2014-01

CONDITIONS: Contraception
Keywords: Pregnancy prevention; Female contraception; Patch
MeSH Terms: interventions — Contraceptives, Oral; Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Gestodene/EE (FC Patch Low, BAY86-5016)
- Arm 2 (Active Comparator)
  Interventions: Drug: Oral contraceptive (equivalent to the active treatment tablets of Levlite), 21-day blister SH D00593A

INTERVENTIONS:
Drug: Gestodene/EE (FC Patch Low, BAY86-5016) — 21-day regimen per cycle (1 patch a week for 3 weeks followed by a 7-day patch-free period) for 7 cycles and placebo tablets matching the conditions of the treatment of Arm 2
  Arms: Arm 1
Drug: Oral contraceptive (equivalent to the active treatment tablets of Levlite), 21-day blister SH D00593A — 21-day regimen per cycle (1 tablet a day for 3 weeks followed by a 7-day tablet-free period) for 7 cycles and placebo patches matching the conditions of the treatment of Arm 1
  Arms: Arm 2

SUMMARY:
Birth Control Patch Study

ELIGIBILITY:
Inclusion Criteria:

* Female subject requesting contraception
* Age: 18 - 45 years (inclusive); smokers must not be older than 35 years at the time of informed consent
* Normal cervical smear not requiring further follow-up (a cervical smear has to be taken at screening visit or a normal result has to be documented within the previous 6 months)
* History of regular cyclic menstrual periods

Exclusion Criteria:

* Pregnancy or lactation
* Significant skin reaction to transdermal preparations or sensitivity to surgical / medical tape
* Any disease that may worsen under hormonal treatment (cardiovascular, liver, metabolic)
* Use of other contraceptive methods than study medication

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 346 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Cycle control parameters and bleeding pattern indices | Treatment cycles 2-7

SECONDARY OUTCOMES:
Number of pregnancies while on treatment up to 14 days after removal of the last patch | 7 treatment cycles each consisting of 28 days and follow-up period of 14 days
Evaluation of blood pressure changes during the dosing-free interval | 7 treatment cycles each consisting of 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (28):
- United States (28):
  - Chandler, Arizona
  - Glendale, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - San Diego, California
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Lake Worth, Florida
  - Leesburg, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Metairie, Louisiana
  - Kalamazoo, Michigan
  - St Louis, Missouri
  - Las Vegas, Nevada
  - New Brunswick, New Jersey
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wexford, Pennsylvania
  - Columbia, South Carolina
  - Richmond, Virginia
  - Renton, Washington
  - Seattle, Washington
  - La Crosse, Wisconsin

REFERENCES:
- [Derived] Merz M, Kroll R, Lynen R, Bangerter K. Bleeding pattern and cycle control of a low-dose transdermal contraceptive patch compared with a combined oral contraceptive: a randomized study. Contraception. 2015 Feb;91(2):113-20. doi: 10.1016/j.contraception.2014.10.004. Epub 2014 Oct 13. PMID 25453585